CLINICAL TRIAL: NCT07132541
Title: Pancreatic Parenchymal Injection of N-Butyl-2-Cyanoacrylate for Pancreaticojejunostomy After Pancreaticoduodenectomy: A Novel Technique
Brief Title: Saleh's Technique for Pancreaticojejunostomy (Pancreatic Parenchymal Injection of N-butyl-2-cyanoacrylate)
Acronym: NBCA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1606/07/2025
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pancreaticoduodenectomy; Postoperative Pancreatic Fistula; Pancreas Cancer; Periampullary Cancer
Keywords: Pancreatic surgery; Anastomotic leak; Tissue adhesive; Postoperative Pancreatic Fistula (POPF); Pancreaticoduodenectomy (PD); Pancreaticojejunostomy (PJ)
MeSH Terms: conditions — Pancreatic Neoplasms; Anastomotic Leak | interventions — Enbucrilate; Tissue Adhesives

STUDY DESIGN:
Intervention Model Description: Patients receiving pancreatic parenchymal injection of N-butyl-2-cyanoacrylate (Histoacryl®) during pancreaticojejunostomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- N-butyl-2-cyanoacrylate (Histoacryl® )Injection Group. (Experimental): Patients in this group will receive pancreatic parenchymal injection of N-butyl-2-cyanoacrylate during pancreaticoduodenectomy.
  Interventions: Drug: Pancreatic parenchymal injection of N-butyl-2-cyanoacrylate(Histoacryl®)

INTERVENTIONS:
Drug: Pancreatic parenchymal injection of N-butyl-2-cyanoacrylate(Histoacryl®) — This procedure is integrated into the standard pancreaticoduodenectomy.
  Injection of Histoacryl® (n-butyl-2-cyanoacrylate) mixed with Lipiodol® (1:1 ratio) into the pancreatic parenchyma circumferentially (3, 6, 9, and 12 o'clock positions) around the main pancreatic duct (MPD) orifice, extending 5-8 mm deep and 5-10 mm laterally from the future anastomotic line, avoiding the main pancreatic duct and vessels. Total volume injected typically ranges from 0.2 ml to 0.6 ml.
  Follow with standard duct-to-mucosa pancreaticojejunostomy:
  * Tying down the posterior duct-to-mucosa sutures.
  * Placing and tying the anterior duct-to-mucosa sutures.
  * Tying down the posterior outer layer sutures.
  * Placing the anterior outer layer sutures. Meticulously avoid glue contact with sutures/mucosa
  Reconstruction: Complete the hepaticojejunostomy and duodenojejunostomy (or gastrojejunostomy).
  Other Names: Histoacryl®, N-butyl-2-cyanoacrylate, Tissue adhesive injection

SUMMARY:
This study investigates the safety and efficacy of injecting N-butyl-2-cyanoacrylate (Histoacryl®) into the pancreatic parenchyma during pancreaticoduodenectomy (PD) to enhance the security of the pancreaticojejunostomy (PJ) anastomosis and reduce postoperative pancreatic fistula (POPF) rates.

DETAILED DESCRIPTION:
Postoperative pancreatic fistula (POPF) remains one of the most significant complications following pancreaticoduodenectomy (PD), with rates ranging from 10% to 30% depending on pancreatic texture and duct size. This study aims to evaluate the use of Histoacryl®, a tissue adhesive, injected into the pancreatic parenchyma to seal leaks and reinforce the anastomotic suture line, particularly in soft pancreases. The study will assess the safety, feasibility, and impact on clinically relevant POPF rates while maintaining exocrine drainage and minimizing parenchymal leakage. Thirty consecutive patients undergoing PD for pancreatic cancer, periampullary cancer, cholangiocarcinoma, or duodenal cancer will be enrolled between July 2025 and July 2026. Preoperative, intraoperative, and postoperative data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy for malignant lesions meeting the curative treatment intent in accordance with clinical guidelines.
* Soft pancreatic texture.
* Small main pancreatic duct diameter (<3 mm).
* Informed consent obtained.

Exclusion Criteria:

* Known hypersensitivity to cyanoacrylate or Lipiodol®.
* Extremely hard, fibrotic pancreas.
* Significant pancreatitis involving the pancreatic remnant.
* Active infection at the surgical site.
* Uncontrolled coagulopathy.
* Unfit patients for surgery due to severe medical illness.
* Inoperable patients with distant metastases, including peritoneal, liver, distant lymph node metastases, and involvement of other organs.
* Irresectable tumors in diagnostic laparoscopy.
* Patients requiring left, central or total pancreatectomy or other palliative surgery.
* Pregnant or breastfeeding women.
* Patients with serious mental disorders.
* Patients with vascular invasion and requiring vascular resection.
* Patients refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pancreatic fistula | 10 days
  A drainage fluid of any measurable volume with an amylase level more than three times the upper normal serum level on or after the 3rd postoperative day.

SECONDARY OUTCOMES:
Incidence of postoperative acute pancreatitis | 1 day post index surgery
  Altered serum amylase count on postoperative day 0 or 1
Incidence of Post-Pancreatectomy Hemorrhage | 90 days
  As defined by the International Study Group for Pancreatic Surgery (ISGPS), grade A, B and C rates
Incidence of intra-abdominal abscess | 90 days
  Collection containing gas bubbles, determining systemic signs of infection
Incidence of biliary fistula | 90 days
  Output of bile from drains on or by post operative day 3
Rate of readmission | 30 days after hospital discharge
  New admission within 30 days of discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Seewald S, Sriram PV, Naga M, Fennerty MB, Boyer J, Oberti F, Soehendra N. Cyanoacrylate glue in gastric variceal bleeding. Endoscopy. 2002 Nov;34(11):926-32. doi: 10.1055/s-2002-35312. No abstract available. PMID 12430080
- [Background] Lamsa T, Jin HT, Sand J, Nordback I. Tissue adhesives and the pancreas: biocompatibility and adhesive properties of 6 preparations. Pancreas. 2008 Apr;36(3):261-6. doi: 10.1097/MPA.0b013e31816714a2. PMID 18362839